CLINICAL TRIAL: NCT01321099
Title: Iron Absorption From Complementary Food Fortificants (CFFs) and Acceptability of CFFs by Beninese Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Federal Institute of Technology (Other)
Collaborators: Université d'Abomey-Calavi (Other)
Responsible Party: Principal Investigator, Prof. Michael B. Zimmermann, Prof, Swiss Federal Institute of Technology
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: CFF_Fe_Study
Record Dates: First submitted 2011-03-22; First posted 2011-03-23 (Estimated); Last update posted 2012-11-08 (Estimated); Status verified 2012-11

CONDITIONS: Iron Deficiency; Anemia
Keywords: Iron absorption; Complementary food fortificant; Young children
MeSH Terms: conditions — Iron Deficiencies; Anemia | interventions — Fe(III)-EDTA; 6-Phytase; Ascorbic Acid

STUDY DESIGN:
Who Masked: Participant

ARMS (3):
- NaFeEDTA (Experimental)
  Interventions: Other: NaFeEDTA
- Phatase (Experimental)
  Interventions: Other: Phytase
- Vitamin C (Experimental)
  Interventions: Other: Vitamin C

INTERVENTIONS:
Other: NaFeEDTA — Labeled iron as FeSO4 or NaFeEDTA added to a test meal
  Arms: NaFeEDTA
Other: Phytase — Labeled iron as FeSO4 added to a test meal with or without phytase and with or without vitamin C
  Arms: Phatase
Other: Vitamin C — Labeled iron as FeSO4 added to a test meal with or without vitamin C
  Arms: Vitamin C

SUMMARY:
Iron deficiency (ID) is still a main public health problem in sub-Saharan Africa. Iron deficient children have an increased risk for anemia which is associated with adverse infant development that might be partly irreversible. In sub-Saharan Africa, the etiology of ID in children is multifactoral; but the major causes are low iron dietary bioavailability and intake from monotonous cereal-based complementary foods. Children < 5 years old can benefit from iron-fortified complementary foods; however, these fortified complementary foods are often not adapted to the requirements of children in specific setting. The investigators developed a complementary food fortificant (CFF) which is added to local porridge and is deemed to meet the nutrient intake requirement for iron in children 1-3 years of age. The CFF is lipid-based and can therefore, if regularly used, increase the daily energy intake of children which is often too low in developing countries with cereal-based diets.

The iron absorption from the mixture of CFF and porridge has to be optimized because it contains quite a high amount of phytate, a well-known inhibitor of iron absorption. To optimize iron absorption the investigators are planning three iron absorption studies using different compounds of iron (FeSO4 + NaFeEDTA), additional vitamin C and phytase, which is able to degrade phytate. In the first study, iron absorption will be determined from a mixture of CFF and porridge fortified with 1) 6 mg FeSO4 and 2) 6 mg FeSO4 plus additional vitamin C. In the second study, the test meals will be fortified with 1) 6 mg FeSO4 and 2) a mixture of 3 mg FeSO4 + 3 mg NaFeEDTA. In the third study, test meals will be fortified with 1) 6 mg FeSO4, 2) 6 mg FeSO4 plus phytase, and 3) 6 mg FeSO4 plus additional vitamin C and phytase. Iron absorption will be determined by incorporation of labeled iron into erythrocytes, 14 days after the administration of a test meal containing labeled iron (stable isotope technique). Sixty apparently healthy Beninese children 12-36 months of age with a body weight > 8.3 kg will be included in the study. Additionally, the investigators will test acceptability of CFFs based on different composition formulas by interviewing the parents/legal guardians of the children after feeding the CFF for a defined period.

The results of these studies will provide important insights to optimize the iron absorption of young children from a CFF mixed with local traditional porridge in developing countries. Furthermore the studies will provide information on the acceptability of CFFs in such a setting.

ELIGIBILITY:
Inclusion Criteria:

* Female or male children, 12 - 36 months of age
* A body weight of at least 8.3 kg; weight for age ≥ -3 Z-score
* No malaria parasites in the blood smear + negative malaria rapid test
* No hematuria
* No intake of mineral/vitamin supplements 2 weeks before and during the study
* No metabolic or gastrointestinal disorders

Exclusion Criteria:

* Fever (body temperature > 37.5 °C)
* Severe anemia (hemoglobin < 8.0 g/dl)
* Regular intake of medication
* Blood transfusion or significant blood loss (accident, surgery) over the past 4 months
* Currently participating in another clinical trial or having participated in another clinical trial during the last 3 months prior to the beginning of this study
* Former participation in a study involving administration of iron stable isotopes
* Subject who cannot be expected to comply with study protocol
* Eating disorders or food allergy

Ages: 12 Months to 36 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2011-05; Primary Completion 2012-06 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Iron isotope ratio in blood samples | Study day 17 (16 days after administration of isotopic label in the first test meal/End of the study)
  Whole blood samples will be collected to measure the shift in iron isotope ratios 16 days after administration of isotopic label in the first test meal.
  First test meal on study day 1, Second test meal on study day 2, Third (last) test meal on study day 3, Measurement of iron isotopic shift in blood samples collected on study day 17

CONTACTS AND LOCATIONS:
Overall Officials: Richard Hurrell, Prof, Principal Investigator — Swiss Federal Institute of Technology (ETH Zürich)
Locations (1):
- University of Abomey-Calavi, Cotonou, Cotonou, Benin